CLINICAL TRIAL: NCT04823156
Title: The Effect of Calcium Intake on Calcium and Bone Metabolism During Load Carriage in Women: a Randomised Controlled Trial
Brief Title: The Effect of Calcium Intake on Calcium and Bone Metabolism During Load Carriage in Women
Acronym: En-Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Army Health Branch, British Army (Other Government)
Collaborators: University of East Anglia (Other); Osteolabs, GEOMAR (Unknown)
Responsible Party: Principal Investigator, Dr. Thomas O'Leary, Higher Scientific Officer, Army Health Branch, British Army
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1021/MODREC/19
Record Dates: First submitted 2020-07-07; First posted 2021-03-30 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Calcium Deficiency
Keywords: Military; Stress Fracture; Calcium; Bone Metabolism
MeSH Terms: conditions — Fractures, Stress | interventions — Calcium

STUDY DESIGN:
Intervention Model Description: Crossover randomised controlled trial.
Masking Description: Calcium supplements will be provided open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Supplementation (Experimental): 1000 mg of calcium carbonate one hour before exercise
  Interventions: Dietary Supplement: Calcium
- No Calcium Supplementation (No Intervention): No calcium supplementation

INTERVENTIONS:
Dietary Supplement: Calcium — Daily calcium food supplement.
  Arms: Calcium Supplementation

SUMMARY:
This randomised trial will investigate the effect of calcium supplementation on bone and calcium metabolism in women during acute load carriage exercise. This study will test the hypothesis that calcium supplementation before load carriage exercise will attenuate the decline in serum ionised calcium and increase in parathyroid hormone and bone resorption.

DETAILED DESCRIPTION:
Endurance exercise decreases serum ionised calcium and increases parathyroid hormone and bone resorption. These disturbances to calcium homeostasis can be attenuated by calcium supplementation before exercise. Military field exercises are characterised by high exercising energy expenditures, restricted dietary intake, and prolonged periods of load carriage. These exercise and nutritional challenges can result in impaired bone turnover, a negative calcium balance, and an increased risk of stress fracture. It is unknown if military load carriage disturbs calcium homeostasis and whether calcium supplementation before exercise can attenuate this disturbance. This crossover randomised controlled trial will investigate the effect of acute calcium supplementation on bone and calcium metabolism in women during acute load carriage exercise. Each participant will complete two 2 h load carriage trials. The trials will be performed after either consuming 1000 mg of calcium one hour before or with no treatment. During each experimental trial blood and urine will be sampled for markers of bone and calcium metabolism.

Primary Outcome: The absolute change in urine calcium balance (Ca44:Ca42) between pre- and post-load carriage will be compared between the non-supplemented (Control) and calcium supplemented trial (Supplement) using one-way ANCOVAs with pre-load carriage calcium balance (either as a ratio, or both the numerator and denominator) as the covariate, or a linear mixed model with the restricted maximum likelihood estimation to allow incorporation of incomplete data.

Secondary Outcomes: Circulating measures of bone turnover and calcium metabolism during load carriage will be compared between Control and Supplement using linear mixed models with the restricted maximum likelihood estimation to allow incorporation of incomplete data.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex;
2. Aged 18 to 36 years old;
3. Maximal rate of oxygen uptake of ≥ 35 ml∙kg-1∙min-1;
4. Weight stable (no change in self-reported body mass ≥ 5% over the previous 3 months);
5. BMI between 18 and 30 kg∙m2;
6. Not pregnant.

Exclusion Criteria:

1. Evidence of disordered eating (≥ 20 on the EAT-26);
2. Self-reported change in body mass of ≥ 5% over the previous 3 months;
3. Vitamin D deficient (total 25(OH)D < 30 nmol∙L-1);
4. Maximal rate of oxygen uptake of < 35 ml∙kg-1∙min-1;
5. Total body BMD T-score of < -1;
6. Evidence of menstrual disturbance (oligomenorrhoea: < 9 menstrual cycles in previous 12 months or amenorrhoea: ≤ 3 menstrual cycles in the previous 12 months);
7. Pregnant;
8. Current smoker, or stopped smoking within the last three months;
9. Taking any medications known to affect bone or calcium metabolism (e.g. treatment for thyroid disorders);
10. Self-declared history of heart, liver or kidney disease, diabetes or thyroid disorder;
11. Self-reported stress fracture or any other bone injuries in the previous 12 months;
12. Anaemia (haemoglobin <12 g∙/dL-1).
13. Currently using the implant, injection, or the progesterone-only pill ('mini pill').

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-05-19 (Estimated); Study Completion 2023-05-19 (Estimated)

PRIMARY OUTCOMES:
Change in calcium balance. | Before and immediately after exercise.
  The ratio of the calcium isotopes Ca44:Ca42 in spot urine samples.

SECONDARY OUTCOMES:
Circulating calcium isotopes during load carriage. | Before and immediately after exercise.
  The ratio of the calcium isotopes Ca44 and Ca42 (Ca44:Ca42) in blood.
Bone turnover during load carriage. | 0, 20, 40, 60, 80, 100, and 120 minutes during, and 15, 30, 60 and 90 minutes following, exercise.
  Circulating concentration of procollagen type 1 N-terminal propeptide (P1NP), beta carboxy-terminal cross-linking telopeptide of type 1 collagen (βCTX), osteocalcin, and sclerostin.
Calcium metabolism during load carriage. | 0, 20, 40, 60, 80, 100, and 120 minutes during, and 15, 30, 60 and 90 minutes following, exercise.
  Circulating concentration of ionized calcium, phosphate, and intact parathyroid hormone.
Dermal calcium loss. | During exercise.
  Concentrations of total calcium and the ratio of the calcium isotopes Ca44 and Ca42 (Ca44:Ca42) in sweat.

OTHER OUTCOMES:
Change in muscle strength during load carriage. | Before and immediately after exercise.
  Loss of muscle strength in the knee extensors and flexors measured by Biodex in response to load carriage exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Army Health and Performance Laboratory, Camberley, Surry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be owned by UK Ministry of Defence, not the Principal Investigator. Data will be made available where possible by the Principal Investigator assuming the appropriate approvals are granted by the UK Ministry of Defence.

REFERENCES:
- [Derived] Coombs CV, Greeves JP, Young CD, Irving AS, Eisenhauer A, Kolevica A, Heuser A, Tang JCY, Fraser WD, O'Leary TJ. The effect of calcium supplementation on bone calcium balance and calcium and bone metabolism during load carriage in women: a randomized controlled crossover trial. J Bone Miner Res. 2025 Jun 3;40(6):753-765. doi: 10.1093/jbmr/zjaf004. PMID 39804018
- [Derived] Coombs CV, Wardle SL, Shroff R, Eisenhauer A, Tang JCY, Fraser WD, Greeves JP, O'Leary TJ. The effect of calcium supplementation on calcium and bone metabolism during load carriage in women: protocol for a randomised controlled crossover trial. BMC Musculoskelet Disord. 2023 Jun 16;24(1):496. doi: 10.1186/s12891-023-06600-w. PMID 37328859